CLINICAL TRIAL: NCT06565429
Title: A Feasibility Study of Delivery of the 5-Step Method Intervention for Family Members of Persons With Substance Use Disorder in the United States
Brief Title: Feasibility of the 5-Step Method in the U.S.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-FY2024-145
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Family Members; Relatives; Substance-Related Disorders; Alcohol-Related Disorders; Coping Skills; Stress, Psychological; Stress Physiology
Keywords: Social Support
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Step Method Intervention Group (Experimental): Receives the 5-Step Method intervention self-help handbook and emails every two weeks to encourage continued use
  Interventions: Behavioral: 5-Step Method Intervention
- Control Group (No Intervention): Standard of care.

INTERVENTIONS:
Behavioral: 5-Step Method Intervention — The 5-Step Method (5SM) intervention is delivered through a self-help handbook: There are writing prompts for the affected family member (AFM) in each step. The steps end with a summary, a space to reflect and a statement that the step is complete but can be reviewed as needed. The steps are: 1.Explore how the relative's drug and/or alcohol misuse is affecting the family member, causing stress and strain. 2.Determine the information the AFM needs to understand the situation using evidence-based websites in the handbook. 3.Reflect on coping styles, and which ones might be useful. 4.Determine who is a source of positive social support, and who could be one that the AFM has not used yet. 5.Review steps 1-4 and determine if the AFM is feeling less stress and strain, or if more help is needed and use websites to look for additional help. The activities should take about 1 hour per week.
  Arms: 5-Step Method Intervention Group

SUMMARY:
The purpose of this study is to see if it is possible (feasible) to introduce a behavioral intervention for family members affected by a relative's misuse of drugs and/or alcohol in the United States. The intervention is called the 5-Step Method. It will be a randomized control trial, with a total of 36 participants, and 18 in each group. The study lasts for approximately 12 weeks for the participant. The intervention group will receive a self-help handbook of the 5-Step Method, and the control group will not. Although the control group will not receive an intervention from the research team, they are allowed to look for and use any currently available program for affected family members (for example, Al-Anon, or Nar-Anon) during the study period. The study is being done because the 5-Step Method has not been used or evaluated in the U.S. (or the creators are unaware that it is in use here). There are two aims (objectives): (1) to see if it is feasible to introduce the 5-Step Method into the U.S.; (2) to look at trends in the baseline and followup survey scores to see if there is evidence of preliminary participant response.

DETAILED DESCRIPTION:
The study will be implemented in the Northern Shenandoah Valley area. A participant in the study will be an affected family member of someone with drug and/or alcohol misuse who has been experiencing stress as a result of the substance misuse for at least the past six months. Both stress and their relative's misuse will be self-identified by the participant. Recruitment for the study will include advertisements via social media, local newspaper notices, and flyers posted at stores and healthcare sites. Once potential participants have contacted the PI and have been screened, consented, and have completed the baseline survey, they will be randomized into either the intervention group or the control group. Once randomized the participant and PI will no longer be blinded to the treatment condition. Those in the intervention group will receive the self-help handbook via the U.S. mail. The control group does not receive an intervention, but could use currently available programs if desired, although information about these programs will not be provided by the PI. All participants will receive emails at regular intervals during their 12-week study period. Because the intervention is completed at the individual level, study recruitment will occur on a rolling basis until 36 participants have been enrolled. Data regarding the feasibility of the study (recruitment, retention, refusal rates, etc.) will be collected. Baseline and follow up surveys will be compared for evidence of participant response.

ELIGIBILITY:
* at least 18 years old
* able to read, write, speak, and understand English
* live in approximately 100-mile radius of Winchester, VA/ in the Northern Shenandoah Valley
* be a family member who self-reports stress/strain because of a relative's drug and/or alcohol misuse
* have access to the Internet and a smartphone or larger device to complete study surveys
* have a personal email address they do not share with others that can receive study related emails
* have the ability to freely consent to participate in the study based on their understanding

Exclusion Criteria:

-if person states the relative with alcohol and/or drug misuse is physically violent towards others

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | One year post completing the intervention
  Scores on Acceptability of Intervention Measure (Weiner et al., 2017), a validated and standardized instrument combined with eight other acceptability questions specific to the 5-Step Method Handbook.
Study process rates | One year post completing the intervention. Rates will be tallied at the end of the study
  Study process rates will be assessed by quantitatively tracking the recruitment rate, retention rate, refusal rate, eligibility rate, and study completion rate.
Likelihood of adverse events | One year post completing the intervention
  Safety will be assessed for all participants by quantitatively summarizing the number of adverse events that are considered to be unexpected, serious, and/or possibly or definitely related to the study
Resources | One year post completing the intervention
  How much time all individual participants spent filling out the surveys, assessed via a survey
Adherence to treatment protocol | 12 weeks after starting study, if placed in the intervention group
  The adherence to treatment protocol will be assessed by asking the intervention group questions about how they interacted with the self-help handbook to determine if they used the handbook as designed or if they used it in some other way.
Marketing | One year post completing the intervention. Will review responses and tally results
  Marketing of the study will be assessed by asking those who inquire about the study where they learned about the study to determine which locations may be better for recruitment in future studies.
Ease of use | One year post completing the intervention
  Ease of use of the study will be assessed by asking participants two questions at the end of the follow-up survey about the way the surveys were worded. The answers of these questions will be reviewed and tallied as well as qualitatively described. The surveys of the study are validated tools, and the only allowed changes to the survey questions were to change from UK English to US English on spelling alone (behaviour to behavior for example). Syntax and word choice were not allowed to be changed. It is possible that how the phrases are stated and the words used will not be as easy to read for an American as compared to someone from the UK, where the intervention was created. The two questions ask if there were any difficulties understanding the survey, and if so, did they think this may have affected how they answered any of the questions.

SECONDARY OUTCOMES:
Stress | Baseline and change over 12 week period
  Family Member Impact Questionnaire (FMI) Scores range from 0-48, with higher scores indicating higher stress.
Coping | Baseline and change over 12 week period
  Symptom Rating Test (SRT) Scores range from 0-90. There are three subscales of coping, with higher scores on two subscales generally associated with higher scores on stress and strain. One subscale is generally associated with lower scores on stress and strain.
Strain | Baseline and change over 12 week period
  Coping Questionnaire (CQ) Scores range from 0-60, higher scores indicating higher scores higher strain.
Social Support | Baseline and change over 12 week period
  Alcohol, Drugs, and the Family Social Support Scale (ADF-SSS) Scores range from 0-75 for the total score. Two subscales with higher scores show improved social support, while the third subscale should have lower numbers when there is an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Therese M Collins, MS, RN, Principal Investigator — Villanova University; Helene Moriarty, PhD, RN, FAAN, Principal Investigator — Villanova University
Locations (1):
- Online Study, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated participant data is planned to be shared

REFERENCES:
- [Background] Copello A, Templeton L, Orford J, Velleman R, Patel A, Moore L, MacLeod J, Godfrey C. The relative efficacy of two levels of a primary care intervention for family members affected by the addiction problem of a close relative: a randomized trial. Addiction. 2009 Jan;104(1):49-58. doi: 10.1111/j.1360-0443.2008.02417.x. PMID 19133888
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Velleman, R., Orford, J., Templeton, L., Copello, A., Patel, A., Moore, L., Macleod, J., & Godfrey, C. (2011). 12-month follow-up after brief interventions in primary care for family members affected by the substance misuse problem of a close relative. Addiction Research & Theory, 19(4), 362-374. https://doi.org/10.3109/16066359.2011.564691
- [Background] Orford, J., Templeton, L., Patel, A., Copello, A., & Velleman, R. (2007a). The 5-step family intervention in primary care: I. strengths and limitations according to family members. Drugs: Education, Prevention and Policy, 14(1), 29-47. https://doi.org/10.1080/09687630600997451